CLINICAL TRIAL: NCT03521895
Title: An Integrated Analysis of the Effectiveness of Intravitreal (IVT) Aflibercept (Eylea) in Routine Clinical Practice Based on Two Large Observational Studies
Acronym: GALAXY
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19694
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment naïve wAMD: Treatment naïve patients with wAMD treated with IVT aflibercept from the two underlying studies PERSEUS and RAINBOW
  Interventions: Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Eylea (Aflibercept, VEGF Trap-Eye, BAY86-5321) — Patients observed with regular and irregular treatment course

SUMMARY:
The aim of this integrated analysis is to describe the effectiveness of Eylea in an integrated pooled analysis using existing individual patient data of two non-interventional studies RAINBOW and PERSEUS.

The primary objective of this integrated analysis is to describe the effectiveness of Eylea on the mean change from baseline in visual acuity (VA) at 12 months in Wet age-related macular degeneration (wAMD) treatment naïve patients.

ELIGIBILITY:
Inclusion Criteria:

PERSEUS

* Patients with wet AMD treated with Eylea (in accordance with the local Summary of Product Characteristics, SPC)
* Documentation of at least one Aflibercept (Eylea) injection
* Assessment of at least one visual acuity measurement with available VA letter score for the study eye at baseline and at least one post-baseline assessment of visual acuity with available VA letter score for the study eye and valid for analysis, i.e. measured at least 5 days after an injection RAINBOW
* Patient with a diagnosis of wet AMD will be enrolled after the decision for treatment with Aflibercept (Eylea) has been made
* Patient who meet the local indication criteria for Eylea treatment
* At least one BCVA after the 1st Eylea injection
* BCVA at baseline
* Patient with no history of retinal disease
* Patient not previously treated with any macular laser or any anti-VEGF intravitreal injections for the study eye (for fellow eye allowed).
* For patients with both eyes treated, the eye firstly treated at initial visit will be considered as study eye. If both eyes are treated during initial visit, the treated eye with worst Best-Corrected Visual Acuity (BCVA) at M0 will be retained. If the two conditions are similar the study eye is the Right eye by convention
* Patient with 1st injection of Eylea from 01 January 2014 until 30 April 2015 will be enrolled Exclusion criteria PERSEUS
* Exclusion criteria as listed in the local SPC
* Scar, fibrosis, or atrophy involving the center of the fovea in the study eye
* All patients previously treated with any macular laser or any anti-VEGF intravitreal injections for the study eye will additionally be excluded for this integrated analysis
* Any concomitant therapy with another agent to treat wet AMD in the study eye RAINBOW
* Patient who does not meet the local indication criteria for Eylea treatment. Contraindications listed in the SmPCs must be taken into account
* Patient with another retinal disease: diabetic retinopathy, diabetic macular oedema (DME), myopic choroidal neovascularization, retinal vein occlusion (RVO), central serous chorioretinopathy (CSC), angioid streaks
* Patient who has previously been treated with any macular laser (laser and/or visudyne/PDT) or any anti-VEGF intravitreal injections for the study eye
* Patient taking part in an interventional study at the time of enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This integrated analysis will include only treatment naïve patients with wAMD treated with IVT aflibercept from the two underlying studies PERSEUS and RAINBOW.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Absolute difference in visual acuity (VA) change from baseline will be calculated for each patient as: VA letter score at month 12 - VA letter score at baseline | At baseline and 12 months

SECONDARY OUTCOMES:
Mean time from diagnosis by the treating physician to start of treatment | At baseline
Proportion of patients gaining 5, 10 or 15 or more letters | At 12 months
Proportion of patients with ≥70 letters VA | At 12 months
Proportion of patients with ≥73 letters VA | At 12 months
Proportion of patients losing 5, 10 or 15 or more letters | At 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

REFERENCES:
- See also: Click here to find results for studies related to Bayer products. — http://clinicaltrials.bayer.com/